CLINICAL TRIAL: NCT02372643
Title: Pilot Interventional Study on Clitoral Ultrasound Measures and Psychobiological Correlates of Female Sexual Function
Brief Title: Ultrasound and Psychobiological Correlates of Female Sexual Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Mario Maggi, Full Professor of Endocrinology, University of Florence
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ANDRO-AOUC-2015-01
Record Dates: First submitted 2015-02-12; First posted 2015-02-26 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Healthy
Keywords: clitoris; sexuality; vascularization; doppler; ultrasound; reference; female; Pilot Projects; Vagina/ultrasonography; Urethra/ultrasonography; Regional Blood Flow/physiology; Arteries/ultrasonography; Clitoris/ultrasonography; Reference values; Clitoris/blood supply
MeSH Terms: conditions — Sexuality; Neovascularization, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sexually healthy women (Other): 20 sexually healthy volunteer women will be enrolled from subjects consulting our outpatient clinic (subjects free from sexual dysfunction). Hormonal and ultrasound parameters and self-administered questionnaires will be evaluated.
  Interventions: Other: clitoral, transvaginal and transrectal ultrasound

INTERVENTIONS:
Other: clitoral, transvaginal and transrectal ultrasound — Doppler Ultrasound assessment of clitoral hemodynamics will be performed in all subjects. Transvaginal and transrectal ultrasound will be performed in subjects giving their consent to these procedures.

SUMMARY:
Monocentric pilot interventional study. The aim of the study is to assess clitoral doppler ultrasonographic parameters in a population of sexually healthy volunteer women in order to obtain reference values. Psychobiological correlates of female sexual function will also be studied through hormonal testing and psychological evaluation.

ELIGIBILITY:
Inclusion Criteria:

* sexually healthy
* evidence of a personally signed and dated informed consent.

Exclusion Criteria:

* any uncontrolled or unstable, acute or chronic disease
* alcohol or drugs abuse
* sexual dysfunction
* any overt psychiatric or psychological condition assessed through psychological evaluation and/or self-administered validated questionnaires.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Clitoral artery peak systolic velocity and acceleration | baseline
  This will not be evaluated in different time frames but evaluated in order to assess reference values in sexually healthy women and compared with subjects with sexual dysfunction.

SECONDARY OUTCOMES:
Female sexual function assessed through the Female Sexual Function Index (FSFI) | baseline
General psychopathology assessed through the Middlesex Hospital Questionnaire (MHQ) | baseline
  See above
Body image is investigated through the Body Uneasiness Test (BUT) | baseline
Measurement of the thickness of the urethrovaginal space | baseline
Measurement of the thickness of the endometrial lining | baseline
Hormonal parameters (17β-estradiol, total testosterone, LH, FSH, TSH, PRL, delta-4-androstenedione, DHEAS, 17-Hydroxyprogesterone, SHBG) | baseline
Metabolic parameters (total cholesterol, HDL, triglycerides, glycemia, insulin, glycated hemoglobin) | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mario Maggi, Principal Investigator — University of Florence
Locations (1):
- Ambulatori di Medicina della Sessualità e Andrologia, Florence, Italy

REFERENCES:
- [Background] Battaglia C, Nappi RE, Mancini F, Cianciosi A, Persico N, Busacchi P, Facchinetti F, de Aloysio D. Menstrual cycle-related morphometric and vascular modifications of the clitoris. J Sex Med. 2008 Dec;5(12):2853-61. doi: 10.1111/j.1743-6109.2008.00972.x. Epub 2008 Aug 28. PMID 18761595
- [Background] Battaglia C, Battaglia B, Mancini F, Nappi RE, Paradisi R, Venturoli S. Moderate alcohol intake, genital vascularization, and sexuality in young, healthy, eumenorrheic women. A pilot study. J Sex Med. 2011 Aug;8(8):2334-43. doi: 10.1111/j.1743-6109.2011.02310.x. Epub 2011 May 19. PMID 21595833
- [Background] Battaglia C, Nappi RE, Mancini F, Alvisi S, Del Forno S, Battaglia B, Venturoli S. PCOS and urethrovaginal space: 3-D volumetric and vascular analysis. J Sex Med. 2010 Aug;7(8):2755-64. doi: 10.1111/j.1743-6109.2009.01651.x. Epub 2010 Jan 6. PMID 20059655